CLINICAL TRIAL: NCT06525896
Title: Research on Effectiveness of Non-surgical Spinal Decompression Therapy and Outcomes With Radiographic Evaluation
Brief Title: Non-surgical Spinal Decompression Therapy and Outcomes
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Stanford University (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY007409: NSSD-RESTORE
Record Dates: First submitted 2024-07-03; First posted 2024-07-29 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain; Herniation, Disc; Sciatic Radiculopathy; Intervertebral Disc Stenosis of Neural Canal; Intervertebral Disc Injury
Keywords: decompression; non-surgical; spine; low back; pain; traction; vertebral axial decompression; spinal traction; stretch; spinal decompression therapy; non-surgical spinal decompression; lumbar; lumbar decompression; back pain treatment; herniated disc therapy; degenerative disc disease treatment; non-invasive spine therapy; chronic back pain relief; Intervertebral Disc Displacement; back pain; lumbar vertebrae; physical therapy modalities; musculoskeletal manipulations; rehabilitation; therapeutics
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Pain; Back Pain | interventions — Traction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NSSD (Experimental): This group will receive non-surgical spinal decompression (20x over 6-8 weeks). Non-surgical spinal decompression is performed by securing the pelvis in a brace and stabilizing the upper torso. The decompression device provides an inferior force along a vector targeting the level of pathology by pulling on the pelvic brace. This causes a comfortable decompression of the spine.
  Interventions: Device: NSSD
- Sham NSSD (Sham Comparator): This group will receive sham non-surgical spinal decompression (20x over 6-8 weeks). Sham non-surgical spinal decompression is performed by securing the pelvis in a brace and stabilizing the upper torso. The decompression device provides an inferior force along a vector targeting the level of pathology by pulling on the pelvic brace, but at a force that does not cause decompression of the spine. This is not perceivable by the participant.
  Interventions: Device: Sham NSSD

INTERVENTIONS:
Device: NSSD — A robotically-controlled distractive force is applied to the lower back to produce decompression of the spinal column.
  Other Names: Vertebral Axial Decompression; Traction
  Arms: NSSD
Device: Sham NSSD — A robotically-controlled distractive force (lower than the intervention) is applied to tension the belt and create a sense of decompression without producing decompression of the spinal column.
  Other Names: Vertebral Axial Decompression; Traction
  Arms: Sham NSSD

SUMMARY:
This project will determine the clinical utility of non-surgical spine decompression for chronic low back pain (LBP). LBP is one of the highest incidence medical conditions that contributes to disability, decreased activities of daily living, decreased quality of life, and inability to work. LBP affects ≈70-85% of people during their lifetime, with ≈20% becoming chronic by age 20-59 years. Many current LBP therapeutics have detrimental long-term effects, undesired side effects, are invasive procedures with low success rates, and do not fare better than conservative care. Further, many chronic musculoskeletal pain patients do not respond to surgery, and many develop dependence on opioids.

This project will implement a small-scale double-blinded, randomized proof-of-concept clinical trial to gather biomechanical and MRI data that will objectively determine the effectiveness of non-surgical spinal decompression (NSSD) over a 12-week longitudinal timeframe. The potential to provide a non-invasive alternative to chronic LBP via NSSD is innovative and addresses the pressing need for safer, more effective pain management options with fewer negative sequelae. NSSD has the potential to greatly improve lives, offering a new paradigm for chronic pain management.

DETAILED DESCRIPTION:
Participants who consent to the study will undergo a comprehensive baseline assessment.

Baseline: During this visit, the patient will receive a chiropractic physician examination that will include reflexes, myotome, dermatome, and orthopedic assessments. If the examination provides evidence of an intervertebral disc pathology and/or sciatica, the patient will be referred to an MRI assessment to confirm diagnosis for standard of care. Based on these assessments, the research team will determine if the participant meets the initial criteria to continue with participation.

Randomization: Participants will be randomized to either non-surgical spinal decompression (20 treatments) or placebo (20 treatments). Participants will not be able to choose the treatment. The participant nor the investigators will know which treatment you are receiving. If a participant receives the placebo treatment, once they are unblinded, they will be able to receive non-surgical spinal decompression should they elect to do so.

Pre-intervention Assessments: Assessments prior to intervention will include 1) 3D motion capture performing functional tasks, 2) electromyography of the lower back and legs, 3) myotonometer tonometry, 4) range of motion, and 5) Sensorimotor reflex measurement. In addition, the participant will complete online questionnaires that include the Defense Veterans Pain Rating Scale 2.0, PROMIS Pain Interference, PROMIS Physical Function, Central Sensitization Inventory, and the Oswestry Disability Index.

Post-intervention Assessments: Assessments after intervention will include 1) 3D motion capture performing functional tasks, 2) electromyography of the lower back and legs, 3) myotonometer tonometry, 4) range of motion, and 5) Sensorimotor reflex measurement. In addition, the participant will complete online questionnaires that include the Defense Veterans Pain Rating Scale 2.0, PROMIS Pain Interference, PROMIS Physical Function, Central Sensitization Inventory, and the Oswestry Disability Index.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of chronic LBP for a minimum of 3 months caused by pathological intervertebral disc, degenerative disc disease, posterior facet syndrome, and/or sciatica.

Exclusion Criteria:

* Known serious spinal pathology (e.g., vertebral fracture, tumor, osteoporosis)
* Evidence of central nervous system involvement of pain
* Other chronic pain conditions
* Pregnancy
* Spinal fusion
* Inability to comply with treatment schedule
* Inability to complete MRIs (e.g., claustrophobia, pacemaker, ferromagnetic implants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Lumbar Spine Magnetic Resonance Imaging (MRI) | Baseline, Pre-Intervention; Immediately after intervention
  Diagnostic imaging of the lumbar spine including T1, T2, and Dixon Fat-Water images. Measures of intervertebral disc height and hydration will be extracted from each lumbar level (L1-L5). Intervertebral disc height will be measured on both T1- and T2-weighted images. The T2-weighted image will assess water signal intensity for intervertebral disc hydration. Muscle quality from the axial Dixon fat-water images will be assessed using the percentage of signal from fat (muscle fat infiltration), a measure of muscle quality. Muscle quality will be assessed in the left and right multifidi, erector spinae, quadratus lumborum, and psoas major muscles.
3D Motion Capture | Baseline, Pre-Intervention; Immediately after intervention
  A markerless motion capture system will measure kinetics and kinematics of functional tasks. Variables of interest include joint angles, limb symmetry, ground reaction forces, double- and single-leg stance percentages, and anticipatory postural acceleration. Tasks include 1) isometric chest raise, 2) tandem balance, 3) sit-to-stand, 4) timed up and go (with gait), and 5) step-up / step-down.
Surface Electromyography | Baseline, Pre-Intervention; Immediately after intervention
  Lumbar neuromotor activation will be assessed with EMG collection (2 kHz) on bilateral musculature, specifically the erector spinae, quadratus lumborum, and gluteus maximus muscles.
Myotonometer | Baseline, Pre-Intervention; Immediately after intervention
  A measure of passive stiffness of the low back muscles (erector spinae, quadratus lumborum, gluteus maximus) at rest (prone) with a MyotonPRO. The MyotonPRO utilizes oscillation accelerometry to measure five output variables of soft tissue: tone (Hz), stiffness (m/sec), elasticity, relaxation (msec), and creep.
Sensorimotor Reflex (H-Reflex) | Baseline, Pre-Intervention; Immediately after intervention
  This electrically evoked response is analogous to a monosynaptic stretch reflex. It is used to assess functionality of the peripheral nervous system (diagnosing and monitoring peripheral neuropathies, radiculopathies, and motor neuron diseases; investigation of mechanisms of motor control, plasticity, and adaptation in response to interventions). The H-reflex is particularly valuable in evaluating the excitability of the alpha motor neurons and their synaptic inputs, which can be affected by IVD lesions.
  A low-intensity electrical stimulus is applied to a mixed peripheral nerve (commonly the tibial nerve) to preferentially activate the Ia afferent fibers. A Digitimer DS7R will provide an electrical stimulus to a sensory neuron. A recording electrode measures the resultant reflexive muscle response which is recorded with surface EMG from the corresponding muscle, providing timing to the sensorimotor reflex loop.

SECONDARY OUTCOMES:
DVPRS 2.0 | Baseline, Pre-Intervention; Throughout trial (approximately 3x/week); Immediately after intervention, 6 months after intervention
  A pain assessment tool that utilizes a numerical rating scale enhanced by functional word descriptors, color coding, and pictorial facial expressions matched to pain levels. Higher scores correlate with increased pain.
PROMIS Physical Function | Baseline, Pre-Intervention; Immediately after intervention, , 6 months after intervention
  A test that measures how well patients with musculoskeletal disorders can perform activities of daily living. High scores correlated with increased function.
PROMIS Pain Interference | Baseline, Pre-Intervention; Immediately after intervention, , 6 months after intervention
  A scale measures how much pain limits a person's ability to participate in physical, mental, cognitive, emotional, recreational, and social activities. Lower scores correlate with increased interference of pain in daily activities.
Oswestry Disability Index | Baseline, Pre-Intervention; Immediately after intervention, 6 months after intervention
  A patient-reported questionnaire for disability associated with the low back that analyzes 10 items. A higher total score correlates with higher disability.
Central Sensitization Inventory | Baseline, Pre-Intervention; Immediately after intervention, 6 months after intervention
  A self-report tool that helps identify patients who may have central sensitization or central sensitivity syndromes. A higher score correlates with higher central sensitization.
International Physical Activity Questionnaire - Short Form | Baseline, Pre-Intervention; Immediately after intervention, 6 months after intervention
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan D Schilaty, DC, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos G, Martin W. Effects of vertebral axial decompression on intradiscal pressure. J Neurosurg. 1994 Sep;81(3):350-3. doi: 10.3171/jns.1994.81.3.0350. PMID 8057141
- [Background] Ramos G. Efficacy of vertebral axial decompression on chronic low back pain: study of dosage regimen. Neurol Res. 2004 Apr;26(3):320-4. doi: 10.1179/016164104225014030. PMID 15142327
- [Background] Gose EE, Naguszewski WK, Naguszewski RK. Vertebral axial decompression therapy for pain associated with herniated or degenerated discs or facet syndrome: an outcome study. Neurol Res. 1998 Apr;20(3):186-90. doi: 10.1080/01616412.1998.11740504. PMID 9583577
- [Background] Macario A, Richmond C, Auster M, Pergolizzi JV. Treatment of 94 outpatients with chronic discogenic low back pain with the DRX9000: a retrospective chart review. Pain Pract. 2008 Jan-Feb;8(1):11-7. doi: 10.1111/j.1533-2500.2007.00167.x. PMID 18211590
- [Background] Karimi N, Akbarov P, Rahnama L. Effects of segmental traction therapy on lumbar disc herniation in patients with acute low back pain measured by magnetic resonance imaging: A single arm clinical trial. J Back Musculoskelet Rehabil. 2017;30(2):247-253. doi: 10.3233/BMR-160741. PMID 27636836
- See also: DRX9000 510(k) approval — https://www.accessdata.fda.gov/cdrh_docs/pdf6/k060735.pdf